CLINICAL TRIAL: NCT00959322
Title: A Prospective Single Center Clinical Study for Capsulotomy Using the LenSx 550 Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LenSx Lasers Inc. (Industry)
Responsible Party: Dr. Melvin Sarayba, M.D., LenSx Lasers, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP-001
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Cataract
Keywords: Capsulotomy
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: LenSx 550 Laser System — Femtosecond laser used to create capsulotomy incision.
  Other Names: LenSx; LenSx 550 Laser; Femtosecond

SUMMARY:
The LenSx 550 laser system is a femtosecond laser intended for use in performing anterior capsulotomy during cataract surgery. The anterior capsulotomy creates a circular opening in the anterior surface of the capsular bag that contains the cataractous crystalline lens. The objective of this study is to evaluate the ability of the LenSx 550 laser to successfully perform anterior capsulotomy during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Must be eligible to undergo cataract extraction by phacoemulsification with primary intraocular lens implantation in at least 1 eye.
* Must be at least 24 years of age.
* Must be willing and able to return for scheduled follow-up examinations.
* Subjects must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* Corneal disease or pathology that precludes applanation of the cornea or transmission of laser wavelength or distortion of laser light.
* Subjects with a poorly dilating pupil or other defect of the pupil that prevents the iris from adequate retraction peripherally are excluded.
* Subjects with residual, recurrent, active ocular or eyelid disease, including any corneal abnormality (for example, recurrent corneal erosion, severe basement membrane disease) in either eye are excluded.
* History of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP>21 mm Hg in either eye.
* Lens/zonular instability such as, but not restricted to, Marfan's Syndrome, Pseudoexfoliation Syndrome, etc.
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye.
* Subjects who are pregnant, lactating, or planning to be pregnant during the course of the study.
* Known sensitivity to planned study concomitant medications.
* Subjects participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.
* Subjects presenting any contraindications to cataract surgery.

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Capsulotomy is complete | 1 day, 1 week, 1 month

SECONDARY OUTCOMES:
No radial tears noted intraoperatively | 1 day, 1 week, 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Kurtz, M.D., Study Chair — LenSx Lasers Inc.; Melvin Sarayba, M.D., Study Director — LenSx Lasers Inc.
Locations (1):
- Semmelweis University, Budapest, Hungary